CLINICAL TRIAL: NCT02571062
Title: A Bioequivalence Study of the Reference Clinical Fexinidazole Tablet vs Proposed Market Formulation in Healthy Male Volunteers of African Sub-Saharan Origin:an Open-label,Randomized,Two-treatment,Single Dose,Replicate Design,Fed Condition
Brief Title: Bioequivalence Study - Reference Clinical Fexinidazole Tablet Versus Proposed Market Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: DNDiHATFEX008
Record Dates: First submitted 2015-06-24; First posted 2015-10-08 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-06

CONDITIONS: Trypanosomiasis, African
Keywords: bioequivalence
MeSH Terms: conditions — Trypanosomiasis, African | interventions — fexinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental formulation (Experimental): crossover design
  Interventions: Drug: Fexinidazole
- final formulation (Experimental): crossover design
  Interventions: Drug: Fexinidazole

INTERVENTIONS:
Drug: Fexinidazole

SUMMARY:
Phase 1 bioequivalence (BE) study. This study is for regulatory purpose to determine BE of the tablet formulation used in the clinical trials and the final marketed tablet formulation under fed condition.

The study will be an open-label, 2-treatment, 2-sequence, 4-period, single-dose, replicate crossover study under fed condition. The 4-period sequences for the replicate design will be TRTR and RTRT, where R designates the reference formulation and T the test formulation. Subject will be allocated randomly to one of the two sequences of treatments according to the randomization list.

DETAILED DESCRIPTION:
Ideally, BE study should be conducted under fasting condition as this is considered to be the most sensitive condition to detect a potential difference between formulations. However as fexinidazole is recommended to be taken with food, as food increased the plasma concentration by 2.5 to 3 fold compared to plasma. BE will be conducted under fed condition, using field adapted meal. The wash-out period should be sufficient to ensure that drug concentrations are below the limit of quantification in all the subjects at the beginning of the next period, a 2 weeks wash-out period will be used. The intra-subject variability of fexinidazole was evaluated based on a previous 3-period cross-over study (1) and was estimated at 25%. As this value was quite high and close to 30%, a replicate design was chosen.

Primary objective:

To assess BE of the clinical trial 600 mg tablet formulation versus (vs.) the proposed market 600 mg tablet formulation of fexinidazole under fed condition after single oral administration of 1200 mg.

Secondary objectives:

To assess the pharmacokinetic profile of the two metabolites fexinidazole sulfoxide and fexinidazole sulfone under the fed condition. To assess the safety and tolerability in healthy volunteers under the same study conditions.

Meal: On each treatment period, fexinidazole will be given with concomitant meal which composition will be as close as possible to field condition

sample size: In order to have 24 evaluable subjects a total of 30 subjects will be recruited in the study.

Study Treatment: Single oral dose of 1200 mg / period :

* Treatment R: Reference formulation, i.e. 2 × 600 mg clinical tablets
* Treatment T: Test formulation, i.e. 2 × 600 mg proposed market tablets

Pharmacokinetic sampling: Pre-dose, and 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 120 and 168 h post-dose Total blood drawn: 390 mL ( Pharmacokinetic = 240 mL + safety = 150 mL)

ELIGIBILITY:
Inclusion Criteria:

1. All subjects to be of sub-Saharan African origins with both parents of sub- Saharan African origins too;
2. Signed ICF;
3. 18 to 45 years old
4. Male subjects with a BMI calculated as weight (kg)/height (m)2 from 18 to 28 kg/m2 at screening
5. Light smokers (less than 5 cigarettes per day, or equivalent e-cigarettes or nicotine patch) or subjects who are non-smokers. No smoking (or use of smoking substitute e.g. nicotine patch) is permitted from screening throughout the study;
6. Normal arterial BP and pulse rate or, if abnormal, considered not clinically significant by the principal Investigator. These will be measured after resting for 5 min;
7. Normal ECG or, if abnormal, considered not clinically significant by the principal Investigator;
8. Registered with the French Social Security in agreement with the French law on biomedical experimentation.

Exclusion Criteria:

1. Who on direct questioning and physical examination have evidence of any clinically significant acute or chronic disease, including known or suspected HIV, HBV or HCV infection
2. With any clinically significant abnormality following review of pre-study laboratory tests (ASAT, ALAT) must be within normal ranges), vital signs, full physical examination and ECG;
3. Who are within the exclusion period defined in the National Register for Healthy Volunteers of the French Ministry of Health;
4. Unwilling to give their informed consent;
5. Who have a positive laboratory test for Hepatitis B surface antigen (HbsAg), or anti-HIV 1/2 or anti- HCV antibodies;
6. Who have a history of allergy, intolerance or photosensitivity to any drug;
7. Who have a history of serious allergy, asthma, allergic skin rash or sensitivity to any drug;
8. Who have a history of HAT;
9. Who are known or suspected alcohol or drug abusers (more than 14 units of alcohol per week, one unit = 8 g or about 10 mL of pure alcohol);
10. Who have a positive alcohol breath test
11. Who drink more than 8 cups daily of beverage containing caffeine;
12. Who have a positive laboratory test for urine drug screening (opiates, cocaine, amphetamine, cannabis, benzodiazepines);
13. Who have undergone surgery or have donated blood within 12 weeks prior to the start of the study;
14. Who have taken any prescribed or over the counter drug (including antacid drug), with the exception of paracetamol (up to 3 g per day) within 2 weeks prior to the first dose administration;
15. Who have already taken fexinidazole;
16. Who have any clinical condition or prior therapy which, in the opinion of the Investigator, made the subject unsuitable for the study;
17. Who participated to any clinical trial with an investigational drug in the past 3 months preceding the first study drug administration.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of fexinidazole following single dose | Pharmacokinetic sampling: Pre-dose, and 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 120 and 168 h
  Area Under the Curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Tarral, MD, Study Director — Drugs for Neglected Diseases
Locations (1):
- Biotrial, Rennes, France